CLINICAL TRIAL: NCT05298449
Title: A Multicenter, Double-blind, Randomized, Parallel, Active-controlled, Phase II Clinical Trial to Evaluate the Efficacy and Safety of HU-045 and Xeomin® in Patients With Moderate to Severe Glabellar Lines
Brief Title: Phase 2 of HU-045 in Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HU-045_P2
Record Dates: First submitted 2022-03-16; First posted 2022-03-28 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Glabellar Lines
Keywords: Glabellar Lines; HU-045; Huons; HuonsBioPharma; Botulinum toxin
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HU-045 group (Experimental): HU-045 Injection group will receive intramuscular injection of HU-045 to a total of 5 glabellar line sites 4 U/0.1ml each.
  HU-045 will be reconstituted from a powder into liquid form by adding 2.5cc of 0.9% sterile saline to the vial, and appropriate volumes will be administered.
  Interventions: Drug: HU-045
- Xeomin® group (Active Comparator): Xeomin® Injection group will receive intramuscular injection of Xeomin® to a total of 5 glabellar line sites 4 U/0.1ml each.
  Xeomin® will be reconstituted from a powder into liquid form by adding 2.5cc of 0.9% sterile saline to the vial, and appropriate volumes will be administered.
  Interventions: Drug: Xeomin®

INTERVENTIONS:
Drug: HU-045 — HU-045 is a medicine that is injected into muscles and used to improve the look of moderate to severe frown lines between the eyebrows (glabellar lines) in adults for a short period of time (temporary). It should be reconstituted with sterile, preservative-free 0.9% saline before use.
  White powder
  Other Names: IncobotulinumtoxinA
  Arms: HU-045 group
Drug: Xeomin® — Xeomin® is a prescription medicine that is injected into muscles and used to improve the look of moderate to severe frown lines between the eyebrows (glabellar lines) in adults for a short period of time (temporary). It should be reconstituted with sterile, preservative-free 0.9% saline before use.
  Other Names: IncobotulinumtoxinA
  Arms: Xeomin® group

SUMMARY:
A Multicenter, Double-blind, Randomized, Parallel, Active-controlled, Phase II Clinical Trial to Evaluate the Efficacy and Safety of HU-045 and Xeomin® in Patients With Moderate to Severe Glabellar Lines

ELIGIBILITY:
Inclusion Criteria:

* 2(Moderate) and/or above of Facial Wrinkle Scale (FWS) score at frown in investigator's live assessment.
* Subject who signed voluntarily in informed consent form and fully understood about this clinical trial.

Exclusion Criteria:

* Subject who has history of any diseases following. (myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis etc.)
* Infection, dermatological condition or scar at the treatment injection sites
* Subject who has marked facial asymmetry
* History of facial nerve palsy or eyebrow/eyelid ptosis
* History of surgical procedures affecting on the lines of forehead and/or middle of the forehead areas
* History of malignant tumor within 5 years (except for basal cell carcinoma
* Any disease and condition that, in the view of the investigator, would interfere with study participation
* Subject who has been treated with any botulinum toxin drug within 6 months
* Subject who takes skeletal muscle relaxants,
* Subject who takes a anticoagulant, antiplatelet, NSAIDs, Vitamin E of over 1,000IU/day (except for low dose aspirin)
* From screening,
* Subject who have positive results of HIV, Syphilis, HBV, HCV
* Drug Hypersensitivity
* Subjects who have hypersensitivity reaction to investigational drug or local anesthetics
* History of Anaphylaxis or severe combined allergy disease
* Subject who has physically untreatable glabellar lines like that can't be spread out even if someone forces it to spread out
* Pregnant and lactating women
* Fertile women and men who have plans to pregnancy and who do not agree to appropriate contraception.
* Participant who has been treated with any investigational drug within 30 days from screening
* Subject who are not eligible for this study based on investigator's judgement.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Percentage of participants whose glabellar lines at maximal frown are improved | Week4
  Investigators will assess participant's glabellar lines with Facial Wrinkle Scale(FWS) at maximal frown; 0=none, 1=mild, 2=moderate or 3=severe.
  Only the participants whose FWS score is 0- or 1-grade when it's assessed and ≥ 2-grade improvement from baseline will be defined as their glabellar lines are improved.

SECONDARY OUTCOMES:
Percentage of participants whose glabellar lines at maximal frown are improved | Week8, Week12
  Investigators will assess participant's glabellar lines with Facial Wrinkle Scale(FWS) at maximal frown; 0=none, 1=mild, 2=moderate or 3=severe.
  Only the participants whose FWS score is 0- or 1-grade when it's assessed and ≥ 2-grade improvement from baseline will be defined as their glabellar lines are improved.
Percentage of participants whose glabellar lines at resting are improved | Week4, Week8, Week12
  Investigators will assess participant's glabellar lines with Facial Wrinkle Scale(FWS) at resting; 0=none, 1=mild, 2=moderate or 3=severe.
  Only the participants whose FWS score is 0- or 1-grade when it's assessed and ≥ 2-grade improvement from baseline will be defined as their glabellar lines are improved.
Subject's satisfaction rate after injection | Week4, Week8, Week12
  Participants will rate their overall satisfaction by answering the question on a Questionnaire using 7-point scale. 6 and/or above grade will be defined as the participant is satisfied about their glabellar lines.
Percentage of subjects who assessed their Glabellar Lines are improved ≥ 2-grade | Week4, Week8, Week12
  Subjects will assess their Galbellar Lines with a 9-point scale from -4 to 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University, Seoul, Dongjak-gu, South Korea